CLINICAL TRIAL: NCT02316509
Title: An Open-Label, Phase I Study of GDC-0927 in Postmenopausal Women With Locally Advanced or Metastatic Estrogen Receptor Positive Breast Cancer
Brief Title: A Study of GDC-0927 in Postmenopausal Women With Locally Advanced or Metastatic Estrogen Receptor Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Seragon Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29656; 2015-000272-95 (EudraCT Number)
Record Dates: First submitted 2014-12-04; First posted 2014-12-15 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

ARMS (2):
- Part I: Dose Escalation - GDC-0927 (Experimental): Participants will receive GDC-0927 orally as a single dose on Day -7. Continuous daily dosing will commence on Day 1. Depending on safety and tolerability, participants will be assigned sequentially to escalating doses of GDC-0927 with use of a standard 3 + 3 design. The starting dose will be 600 milligrams per day (mg/day), followed by dose escalation in 400 milligrams (mg) increments.
  Interventions: Drug: GDC-0927
- Part II: Dose Expansion - GDC-0927 (Experimental): Participants in the expansion cohorts will receive GDC-0927 at MTD/RP2D starting from Day 1 of Cycle 1 (cycle length: 28 days) up to disease progression, unacceptable toxicity, participant withdrawal of consent or study termination.
  Interventions: Drug: GDC-0927

INTERVENTIONS:
Drug: GDC-0927 — GDC-0927 will be administered as per schedule specified in the respective arm.
  Other Names: RO7056119

SUMMARY:
This is an open-label, dose-finding, safety, pharmacokinetics (PK), and evidence-of-activity study of GDC-0927 in postmenopausal women with locally advanced or metastatic Estrogen Receptor Positive (ER+) Human Epidermal Growth Factor Receptor 2 (HER2) breast cancer. The study will be conducted in two parts: Dose escalation and Dose expansion. During dose escalation, GDC-0927 will be administered orally as a single dose on Day -7 for PK evaluation during the lead-in period. Depending on safety and tolerability, participants will be assigned sequentially to escalating doses of GDC-0927 using standard 3+3 design. During dose expansion, there will be no PK week lead-in period. All participants will be treated until disease progression, unacceptable toxicity, participant withdrawal of consent or study termination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of adenocarcinoma of the breast with evidence of either locally recurrent disease not amenable to resection or radiation therapy with curative intent, or metastatic disease, both progressing after at least 6 months of hormonal therapy for ER+ breast cancer
* ER-positive tumor, HER2-negative breast cancer
* No prior treatment with GDC-0810 (allowed only during dose expansion stage)
* No more than 2 prior chemotherapies in the advanced or metastatic setting
* At least 2 months must have elapsed from the use of tamoxifen
* At least 6 months must have elapsed from the use of fulvestrant
* At least 2 weeks must have elapsed from the use of any other endocrine therapy
* At least 3 weeks must have elapsed from the use of any chemotherapy
* Females, 18 years of age or older
* Postmenopausal status as defined by the protocol
* Eastern Cooperative Oncology Group (ECOG) Performance status less than or equal to (</=) 2 (for dose-escalation part) and 0 or 1 (for dose-expansion part)
* Adequate organ function

Exclusion Criteria:

* Untreated or symptomatic brain metastases
* Current treatment with any systemic anti-cancer therapies for advanced disease or any systemic experimental treatment on another clinical trial
* Any of the following within 12 months prior to enrollment: myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of Grade greater than or equal to (>/=) 2, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, or cerebrovascular accident including transient ischemic attack
* Active inflammatory bowel disease or chronic diarrhea, short bowel syndrome, or upper gastrointestinal surgery including gastric resection
* Known Human Immunodeficiency Virus (HIV) infection
* Major surgery within 4 weeks prior to enrollment
* Radiation therapy within 2 weeks prior to enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD)/Recommended Phase II Dose (RP2D) of GDC-0927 | Day-7 through Cycle 1 (cycle length: 28 days)
Percentage of Participants With Adverse Events (AEs) | From screening up to approximately 3 years

SECONDARY OUTCOMES:
Percentage of Participants With Objective Response Assessed by Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) | At screening, every 8 weeks from Cycle 1 (each cycle: 28 days) up to end of treatment (up to approximately 3 years)
Percentage of Participants With Clinical Benefit Assessed by RECIST v1.1 | At screening, every 8 weeks from Cycle 1 (each cycle: 28 days) up to end of treatment (up to approximately 3 years)
Part I: Maximum Observed Plasma Concentration (Cmax) of GDC-0927 | Pre-dose (0 hour [hr]), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24 hrs post-dose on Day -7; Days -5, -4, -3; pre-dose (0 hr) on Day 1 Cycle 1; pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-dose on Day 1 Cycle 2 (cycle length: 28 days)
Part II: Cmax of GDC-0927 | Pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24 hrs post-dose on Day 1 Cycle 1; pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-dose on Day 1 Cycle 2 (each cycle: 28 days)
Part I: Time to Reach Cmax (Tmax) of GDC-0927 | Pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24 hrs post-dose on Day -7; Days -5, -4, -3; pre-dose (0 hr) on Day 1 Cycle 1; pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-dose on Day 1 Cycle 2 (cycle length: 28 days)
Part II: Tmax of GDC-0927 | Pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24 hrs post-dose on Day 1 Cycle 1; pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-dose on Day 1 Cycle 2 (each cycle: 28 days)
Part I: Area Under the Plasma Concentration Versus Time Curve (AUC) of GDC-0927 | Pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24 hrs post-dose on Day -7; Days -5, -4, -3; pre-dose (0 hr) on Day 1 Cycle 1; pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-dose on Day 1 Cycle 2 (cycle length: 28 days)
Part II: AUC of GDC-0927 | Pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24 hrs post-dose on Day 1 Cycle 1; pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8 hrs post-dose on Day 1 Cycle 2 (each cycle: 28 days)
Plasma Half-Life (t1/2) of GDC-0927 | Pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24 hrs post-dose on Day -7; Days -5, -4, -3; pre-dose (0 hr) on Day 1 Cycle 1 (cycle length: 28 days)
Part II: t1/2 of GDC-0927 | Pre-dose (0 hr), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24 hrs post-dose on Day 1 Cycle 1 (each cycle: 28 days)
Part I: Change From Baseline in Corrected QT (QTc) Interval Using Fridericia's Formula, as Assessed by Electrocardiogram (ECG) | Screening (baseline); Days -7, -5, -4, -3; Cycle 2 Day 1; end of treatment (up to approximately 3 years) (each cycle = 28 days)
Part II: Change From Baseline in QTc Interval Using Fridericia's Formula, as Assessed by ECG | Screening (baseline); Cycle 1 Day 1; Cycle 2 Day 1; end of treatment (up to approximately 3 years) (each cycle = 28 days)
Part I: Change From Baseline in RR Interval, as Assessed by ECG | Screening (baseline); Days -7, -5, -4, -3; Cycle 2 Day 1; end of treatment (up to approximately 3 years) (each cycle = 28 days)
Part II: Change From Baseline in RR Interval, as Assessed by ECG | Screening (baseline); Cycle 1 Day 1; Cycle 2 Day 1; end of treatment (up to approximately 3 years) (each cycle = 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (5):
  - Massachusetts General Hospital., Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Cancer Center, Germantown, Tennessee
  - Vanderbilt Ingram Cancer Ctr, Nashville, Tennessee
- Spain (8):
  - ICO I Hospitalet Hospital Duran i Reynals Instituto Catalan de Oncologia de Hospitalet ICO, L'Hospitalet de Llobregat, Barcelona
  - Onkologikoa - Kutxaren Institutu Onkologikoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - MD Anderson Cancer Center Madrid - España; Servicio de Farmacia, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - HM Sanchinarro - CIOCC, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia